CLINICAL TRIAL: NCT05435443
Title: Comparison of Two Respiratory Physiotherapy Treatments in Postcovid-19 Patients. Randomiced Clinical Trial
Brief Title: Comparison of Two Respiratory Physiotherapy Treatments in Postcovid-19 Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, Principal Investigator, Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 260322
Record Dates: First submitted 2022-06-26; First posted 2022-06-28 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: COVID-19; Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the PowerBreathe and PEP Therosold tools group (Experimental)
  Interventions: Device: PowerBreathe and PEP Therosold tools
- perform diaphragmatic breathing, series of abdominal crunches and expiratory exercises group. (Active Comparator)
  Interventions: Device: PowerBreathe and PEP Therosold tools

INTERVENTIONS:
Device: PowerBreathe and PEP Therosold tools — Initially, the following data were collected from each subject in addition to basic epidemiological data:
  M-mode diaphragmatic excursion measurements, both in inspiration and expiration via ultrasound; spirometry is also carried out, obtaining values of forced vital capacity (FVC or FVC), forced expiratory volume (FEV), portion of FVC (FEV1/FVC), peak expiratory flow (PEF), mean expiratory flow, peak inspiratory pressure (PIM) and peak expiratory pressure (PEM). A 30-day treatment plan was carried out in which one group (Tool Group) had to perform 5 minutes of exercise with each tool, alternating with one minute of rest between each minute of exercise, starting with the Therosold PEP® and then the PowerBreathe®. The resistances applied to the devices were marked according to the specific assessment of each subject, in relation to the spirometric values of PIM and PEM.

SUMMARY:
To test the effectiveness of a respiratory physiotherapy treatment plan in patients who have passed COVID-19, comparing two randomized groups, for the performance of different respiratory musculature training protocols. To objectify the results data obtained by means of ultrasound measurements and spirometry, observing the differences obtained at the beginning and end of the study, verifying the effectiveness of the PowerBreathe® ,Therosold PEP® tools and the effectiveness of diaphragmatic, abdominal and expiratory exercises.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Covid and suffering from functional limitations in the respiratory system.
* Patients over 18 years of age.
* Patients under 65 years of age.
* Patientes with cognitive ability to perform spirometry.
* Patients with the physical capacity to perform spirometry

Exclusion Criteria:

* - Patients diagnosed with Covid and without functional limitations in the respiratory system.
* Patients under 18 years of age.
* Patients over 65 years of age.
* Patients without cognitive capacity to perform spirometry.
* Patients without physical capacity to perform spirometry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
peak inspiratory pressure (PIM) | 1 month
  0 miminum ,200 maximum
peak expiratory pressure | 1 month
  0 miminum ,200 maximum
forced vital capacity | 1 month
  0 miminum ,200 maximum

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica de Ávila, Ávila, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gosselink R, Bott J, Johnson M, Dean E, Nava S, Norrenberg M, Schonhofer B, Stiller K, van de Leur H, Vincent JL. Physiotherapy for adult patients with critical illness: recommendations of the European Respiratory Society and European Society of Intensive Care Medicine Task Force on Physiotherapy for Critically Ill Patients. Intensive Care Med. 2008 Jul;34(7):1188-99. doi: 10.1007/s00134-008-1026-7. Epub 2008 Feb 19. PMID 18283429
- [Result] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Result] Lazzeri M, Lanza A, Bellini R, Bellofiore A, Cecchetto S, Colombo A, D'Abrosca F, Del Monaco C, Gaudiello G, Paneroni M, Privitera E, Retucci M, Rossi V, Santambrogio M, Sommariva M, Frigerio P. Respiratory physiotherapy in patients with COVID-19 infection in acute setting: a Position Paper of the Italian Association of Respiratory Physiotherapists (ARIR). Monaldi Arch Chest Dis. 2020 Mar 26;90(1). doi: 10.4081/monaldi.2020.1285. PMID 32236089
- [Result] Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species Severe acute respiratory syndrome-related coronavirus: classifying 2019-nCoV and naming it SARS-CoV-2. Nat Microbiol. 2020 Apr;5(4):536-544. doi: 10.1038/s41564-020-0695-z. Epub 2020 Mar 2. PMID 32123347
- [Result] Pal M, Berhanu G, Desalegn C, Kandi V. Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2): An Update. Cureus. 2020 Mar 26;12(3):e7423. doi: 10.7759/cureus.7423. PMID 32337143
- [Derived] Sanchez-Mila Z, Abuin-Porras V, Romero-Morales C, Almazan-Polo J, Velazquez Saornil J. Effectiveness of a respiratory rehabilitation program including an inspiration training device versus traditional respiratory rehabilitation: a randomized controlled trial. PeerJ. 2023 Dec 15;11:e16360. doi: 10.7717/peerj.16360. eCollection 2023. PMID 38111659